CLINICAL TRIAL: NCT00738751
Title: Phase I Study of LBH589 in Combination With Erlotinib for Advanced Aerodigestive Tract Cancers (CLBH5889CUS11T)
Brief Title: Phase I Study of LBH589 & Erlotinib for Advanced Aerodigestive Tract Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Genentech, Inc. (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15461; LBH589 (Other: Novartis)
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Lung Cancer; Head and Neck Cancer
Keywords: NSCLC; Metastatic; erlotinib; aerodigestive tract cancers; non-small cell lung cancer; H&N cancer
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — Panobinostat; Histone Deacetylase Inhibitors; Erlotinib Hydrochloride; Quinazolines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation Followed by Expansion (Experimental): Eligible participants were enrolled in a 3+3 dose-escalation design to determine the maximum tolerated dose (MTD) of twice weekly panobinostat plus daily erlotinib at 4 planned dose levels (DLs).
  Interventions: Drug: Panobinostat (LBH589); Drug: erlotinib

INTERVENTIONS:
Drug: Panobinostat (LBH589) — Panobinostat was taken twice weekly, for 2 out of 3 weeks of each cycle. Each cycle was defined as a 21-day period. Four dose levels of panobinostat in combination with erlotinib were planned: 1) dose level 1 (DL1) = panobinostat 20 mg by mouth (PO) twice weekly for 2 out of 3 weeks + erlotinib 100 mg PO daily; 2) dose level 2 (DL2) = panobinostat 30 mg and erlotinib 100 mg; 3) dose level 3 (DL3) = panobinostat 30 mg and erlotinib 150 mg; and 4) dose level 4 (DL4) = panobinostat 40 mg and erlotinib 150 mg. Doses were not escalated over the course of treatment of an individual participant.
  Other Names: histone deacetylase inhibitor; HDAC
Drug: erlotinib — Erlotinib was taken daily without interruption. Each cycle was defined as a 21-day period. Panobinostat was taken twice weekly, for 2 out of 3 weeks of each cycle. Four dose levels of panobinostat in combination with erlotinib were planned: 1) dose level 1 (DL1) = panobinostat 20 mg by mouth (PO) twice weekly for 2 out of 3 weeks + erlotinib 100 mg PO daily; 2) dose level 2 (DL2) = panobinostat 30 mg and erlotinib 100 mg; 3) dose level 3 (DL3) = panobinostat 30 mg and erlotinib 150 mg; and 4) dose level 4 (DL4) = panobinostat 40 mg and erlotinib 150 mg. Doses were not escalated over the course of treatment of an individual participant.
  Other Names: Tarceva; quinazoline

SUMMARY:
The main purpose of the study is to:

* Determine the safety and tolerability of erlotinib and LBH589B.
* Establish a recommended phase II expansion dosing of LBH589B and erlotinib in patients with advanced aerodigestive tract cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented diagnosis of advanced/metastatic NSCLC or Head and Neck cancer.
* Male or female patients aged ≥ 18 years old
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Have progressive and measurable disease that can be measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Patients must have discontinued prior systemic chemotherapy by 14 days.
* Patients must meet the following laboratory criteria:

  1. Serum albumin ≥ 3g/dL
  2. Aspartic transaminase (AST/SGOT) and alanine transaminase (ALT/SGPT) ≤ 2.5 x upper limit of normal (ULN)or ≤ 5.0 x ULN if the transaminase elevation is due to leukemic involvement
  3. Serum bilirubin ≤ 1.5 x ULN
  4. Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 ml/min
  5. Serum potassium ≥ lower limit of normal (LLN) and ≤ ULN
  6. Serum phosphorous ≥ LLN
  7. Serum total calcium (corrected for serum albumin) or serum ionized calcium ≥ LLN
  8. Serum magnesium ≥ LLN
  9. Absolute neutrophil count (ANC) (ANC: segmented and bands) ≥ 1.5 X10^9/L
  10. Platelets ≥ 100 X 10^9/L
* Baseline multiple gated acquisition imaging (MUGA) or echocardiogram (ECHO) must demonstrate left ventricular ejection fraction (LVEF) ≥ the lower limit of the institutional normal
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
* Reproductive potential must be either terminated (by surgery, radiation, or menopause) or attenuated by the use of an approved contraceptive method during and for 3 to 6 months following the study.
* Patient instructed that intravenous (IV) bisphosphonates will be withheld for the first 8 weeks of LBH589 therapy due to risk of hypocalcemia.

Exclusion Criteria:

* Impaired cardiac function including any one of the following:

  1. Screening electrocardiogram (ECG) with a corrected QT (QTc) > 450 msec confirmed by central laboratory prior to enrollment to the study
  2. Patients with congenital long QT syndrome
  3. History of sustained ventricular tachycardia
  4. Any history of ventricular fibrillation or torsades de pointes
  5. Bradycardia defined as heart rate < 50 beats per minute. Patients with a pacemaker and heart rate ≥ 50 beats per minute are eligible.
  6. Patients with a myocardial infarction or unstable angina within 6 months of study entry
  7. Congestive heart failure - New York Heart Association (NYHA) class III or IV
  8. Right bundle branch block and left anterior hemiblock (bifascicular block)
  9. Patients with a history of uncontrolled or chronic atrial fibrillation.
* Uncontrolled hypertension, blood pressure (BP) >180/110 on 3 separate occasions despite oral antihypertensive medications
* Concomitant use of drugs with a risk of causing torsades de pointes Concomitant use of CYP3A4 inhibitors
* Patients with documented central nervous system or leptomeningeal metastasis (brain metastasis) at the time of study entry. Patients with prior brain metastasis may be considered if they have completed their treatment for brain metastasis, no longer require corticosteroids, and are asymptomatic.
* Patients with unresolved diarrhea > Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
* Other concurrent severe and/or uncontrolled medical conditions
* Patients who have received chemotherapy < 14 days, any investigational drug < 14 days or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Concomitant use of any anti-cancer therapy (except erlotinib) or radiation therapy.
* Female patients who are pregnant or breast feeding or patients of reproductive potential not using two effective methods of birth control. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of oral LBH589
* Male patients whose sexual partners are WOCBP not using effective birth control
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
* Patients who are not willing to refrain from wearing contact lenses during study participation will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-11; Primary Completion 2013-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 4 Months
  Determine safety and tolerability of erlotinib and LBH589B and establish a recommended phase II expansion dosing of LBH589B and erlotinib in patients with advanced aerodigestive tract cancers.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 48 months
  DCR: The percentage of patients with advanced or metastatic cancer who have achieved complete response (CR), partial response (PR) and stable disease (SD) to a therapeutic intervention in clinical trials of anticancer agents. CR: is defined as disappearance of all target lesions. PR: is defined as at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD. SD: is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since the treatment started.
Progression Free Survival (PFS) by Cancer Type | Up to 48 months
  Progressive Disease (PD) is defined as at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Overall Survival (OS) by Cancer Type | Up to 48 months
  Overall survival (OS) is the duration from date of randomization to date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle Gray, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States